CLINICAL TRIAL: NCT05037474
Title: Contemporary Mechanical Lead Extraction Outcomes From a High-volume Center: Patient Characteristics, Procedural Characteristics and Outcomes.
Brief Title: Contemporary Transvenous Lead Extraction Outcomes
Acronym: TLE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-025
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-08

CONDITIONS: Pacemaker Lead Dysfunction; Pacemaker Electrode Infection; ICD; Endocarditis Infective
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TLE group — all patients underwent a transvenous lead extraction/explantation (TLE) procedure

SUMMARY:
Presentation of procedural safety and outcomes data from a high volume TLE centre

DETAILED DESCRIPTION:
Transvenous lead extraction is crucial procedure in the longterm management of patients with implanted pacemakers or cardioverter defibrillators.

Our study presents the patient and procedural characteristics as well as the outcome data of a cohort undergoing transvenous lead extraction (TLE) with olny mechanical extraction tools at a high-volume TLE centre.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a lead removal procedure

Exclusion Criteria:

* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a lead extractions or lead explantation (defined by the EHRA consensus statement) procedure were prospectively enrolled in the database,
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete or clinical successful lead removal | acute setting (during the surgical procedure)
  Removal of a lead or retention of a part less than 4cm
Percentage of patients undergoing TLE with major and minor complication | acute setting (during the surgical procedure)
  procedure related major and minor complications

SECONDARY OUTCOMES:
long term outcome | >12months follow up
  survival after TLE
Percentage of patients encountering a major or minor sedation complication during TLE | acute setting (during the surgical procedure)
  Complication of cardiologist-directed sedation during TLE procedures

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Lennerz, MD, Principal Investigator — German Heart Center
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany